CLINICAL TRIAL: NCT05014217
Title: Comparaison d'Une thérapie basée Sur la Mentalisation et d'un Traitement inspiré de la thérapie Comportementale Dialectique Sur l'Utilisation Des Services et Sur le Taux d'Abandon Dans Une Population Clinique Adulte Atteinte d'un Trouble de la personnalité du Groupe B
Brief Title: Comparing Mentalization-based Treatment And A Dialectical Behavior Therapy-inspired Treatment On The Utilization Of Services And The Dropout Rate In A Clinical Adult Population With A Cluster B Personality Disorder
Status: Completed | Type: Observational
Sponsor: Ciusss de L'Est de l'Île de Montréal (Other)
Responsible Party: Sponsor
Other Study IDs: STRP1 2020-2193
Record Dates: First submitted 2021-08-13; First posted 2021-08-20 (Actual); Last update posted 2021-10-13 (Actual); Status verified 2021-08

CONDITIONS: Cluster B Personality Disorder (Diagnosis); Borderline Personality Disorder
Keywords: cluster B personality disorder; mentalization-based treatment; dialectical behavior therapy; borderline personality disorder; service utilization; dropout rate; naturalistic study
MeSH Terms: conditions — Disease; Borderline Personality Disorder | interventions — Mentalization-Based Therapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Mentalization-based Treatment: Participants who have been oriented to the mentalization-based treatment among the clinical adult population with a cluster B personality disorder.
  Interventions: Behavioral: Mentalization-based Treatment
- Dialectical Behavior Therapy-inspired Treatment: Participants who have been oriented to the dialectical behavior therapy-inspired treatment among the clinical adult population with a cluster B personality disorder.
  Interventions: Behavioral: Dialectical Behavior Therapy-inspired Treatment

INTERVENTIONS:
Behavioral: Mentalization-based Treatment — An empirically-validated intervention for personality disorders based on the attachment theory and on knowledge from developmental psychology and cognitive neuroscience (Bateman and Fonagy, 2004). Patients assist psychoeducative group meetings beforehand, along with a pretreatment of four to six individual meetings (over four to eight weeks), followed by bi-weekly individual follow-ups and weekly group follow-ups. The treatment lasts two years. Patients have an assessment meeting with their individual therapist and one of the group therapists at the end of each session. Psychiatric follow-up appointments are on an as-needed basis and every patient has a treatment contract with specific and measurable treatment objectives.
  Groups: Mentalization-based Treatment
Behavioral: Dialectical Behavior Therapy-inspired Treatment — A psychotherapy developed by M. Linehan for patients with borderline personality disorder that combines cognitive behavioral therapy techniques (emotional regulation, practical exercises) with Buddhist meditation principles (stress tolerance, acceptance, open-mindedness) (Linehan, M. M. & Dimeff, L., 2001). As opposed to Linehan's model, individual meetings are bi-weekly, no emergency phone service is offered, the mindful meditation module is reorganized into life habits modules, and every module includes mindfulness exercises. Patients assist psychoeducative group meetings beforehand, along with a pre-treatment of 4-6 individual meetings (over 4-8 weeks), followed by bi-weekly individual follow-ups and weekly group follow-ups. The treatment lasts one year, but can be extended to two years for eligible patients who are interested. Psychiatric follow-up appointments are on an as-needed basis. Every every patient has a treatment contract with specific and measurable treatment objectives.
  Groups: Dialectical Behavior Therapy-inspired Treatment

SUMMARY:
Cluster B personality disorders (borderline, narcissistic, antisocial and/or histrionic) are an important clinical consideration because of their high prevalence and associated morbidity. Although many studies examine borderline personality disorder, few of them explore cluster B personality disorders as a whole. In clinical practice, personality disorders are frequently comorbid. Patients who receive services in specialized clinics for these disorders often have a complex diagnosis that include many cluster B personality disorders. Therefore, our study globally examines patients with cluster B personality disorders even though borderline personality disorder is empirically the most studied psychopathology. Previous data suggests that borderline personality disorder has a prevalence of 2% in the general population, of 25% in the clinical psychiatric population and of 15% in all visits to the emergency room. Furthermore, it is associated with social costs estimated from 15,000$ to 50,000$ USD per patient per year. In Quebec, this psychopathology is associated with an increased mortality rate compared to the general population, totaling a loss of nine years for women and 13 years for men of life expectancy. Other studies suggest that borderline personality disorder is often comorbid with other personality disorders, including those in cluster B. The population with comorbid personality disorders have a worse prognosis and a lower chance of reaching symptomatic remission, which is the reason why it is crucial to better understand and study patients with cluster B personality disorders.

The study compares the effectiveness of two psychotherapies for borderline personality disorder, mentalization-based therapy and a modified version of Linehan's dialectical behavior therapy, in a retrospective naturalistic study of patients with at least one cluster B personality disorder who have undergone either treatment. The scarcity of data on cluster B personality disorders and on the comparison between MBT and DBT further highlights the necessity of a naturalistic study like ours to examine both aspects and bring research closer to the clinical setting. Based on clinical observations, the investigators believe that there will be no statistically significant difference between either treatment.

ELIGIBILITY:
Inclusion Criteria:

* Meet the general criteria for a personality disorder
* Be diagnosed with at least one cluster B personality disorder
* Be admitted to the Service of personality and relational disorders and referred to mentalization-based treatment or a treatment inspired from dialectical behavior therapy

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients diagnosed with at least one cluster B personality disorder and admitted to the Service of personality and relational disorders at the Institut universitaire de Santé Mentale de Montréal after being referred to the program and oriented to mentalization-based treatment or dialectical behavior therapy. Patients with comorbid personality disorders are also included to better represent clinical practice.
Sampling Method: Non-Probability Sample
Enrollment: 403 (Actual)
Dates: Start 2015-01-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2021-08-04 (Actual)

PRIMARY OUTCOMES:
Number of Visits To The Emergency Room | One year before the index date (first group therapy meeting) to one year after the index date.
  A comparison of the difference between a patient's number of visits to the emergency room in the year prior to and the year following the index date for each treatment.
Number of Hospitalizations | One year before the index date (first group therapy meeting) to one year after the index date.
  A comparison of the difference between a patient's number of hospitalizations in the year prior to and the year following the index date for each treatment.

SECONDARY OUTCOMES:
Dropout rate | From the beginning until the end of the psychotherapy treatment.
  The comparison of the dropout rate between mentalization-based treatment and dialectical behavior therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Simon Poirier, MD, Principal Investigator — Ciusss de L'Est de l'Île de Montréal

IPD SHARING:
Plan to Share IPD: No
Patients have not consented to have their data be available to researchers outside the institution.

REFERENCES:
- [Background] Ansell EB, Sanislow CA, McGlashan TH, Grilo CM. Psychosocial impairment and treatment utilization by patients with borderline personality disorder, other personality disorders, mood and anxiety disorders, and a healthy comparison group. Compr Psychiatry. 2007 Jul-Aug;48(4):329-36. doi: 10.1016/j.comppsych.2007.02.001. Epub 2007 Apr 6. PMID 17560953
- [Background] Barnicot K, Crawford M. Dialectical behaviour therapy v. mentalisation-based therapy for borderline personality disorder. Psychol Med. 2019 Sep;49(12):2060-2068. doi: 10.1017/S0033291718002878. Epub 2018 Oct 10. PMID 30303061
- [Background] Bateman, A. & Fonagy, P. (2004). Psychotherapy of Borderline Personality Disorder:mentalisation-based treatment. Oxford, UK: Oxford University Press.
- [Background] Bender DS, Dolan RT, Skodol AE, Sanislow CA, Dyck IR, McGlashan TH, Shea MT, Zanarini MC, Oldham JM, Gunderson JG. Treatment utilization by patients with personality disorders. Am J Psychiatry. 2001 Feb;158(2):295-302. doi: 10.1176/appi.ajp.158.2.295. PMID 11156814
- [Background] Cailhol, L., et al. (2015). Surveillance des troubles de la personnalité au Québec : prévalence, mortalité et profil d'utilisation des services, INSPQ (Institut National de santé publique du Québec).
- [Background] Cristea IA, Gentili C, Cotet CD, Palomba D, Barbui C, Cuijpers P. Efficacy of Psychotherapies for Borderline Personality Disorder: A Systematic Review and Meta-analysis. JAMA Psychiatry. 2017 Apr 1;74(4):319-328. doi: 10.1001/jamapsychiatry.2016.4287. PMID 28249086
- [Background] Duggan, C., Huband, N., Smailagic, N., Ferriter, M., & Adams, C. (2007). The use of psychological treatments for people with personality disorder: A systematic review of randomized controlled trials. Personality and Mental Health, 1, 95-125.
- [Background] Linehan, M. M. & Dimeff, L. (2001). Dialectical Behavior Therapy in a nutshell [archive], The California Psychologist, 34, 10-13.
- [Background] Linehan MM, Comtois KA, Murray AM, Brown MZ, Gallop RJ, Heard HL, Korslund KE, Tutek DA, Reynolds SK, Lindenboim N. Two-year randomized controlled trial and follow-up of dialectical behavior therapy vs therapy by experts for suicidal behaviors and borderline personality disorder. Arch Gen Psychiatry. 2006 Jul;63(7):757-66. doi: 10.1001/archpsyc.63.7.757. PMID 16818865
- [Background] Links PS, Heslegrave R, van Reekum R. Prospective follow-up study of borderline personality disorder: prognosis, prediction of outcome, and Axis II comorbidity. Can J Psychiatry. 1998 Apr;43(3):265-70. doi: 10.1177/070674379804300305. PMID 9561315
- [Background] Luyten P, Leichsenring F, Abbass A, Hilsenroth M, Rabung S, Steinert C. What to conclude from a non-randomized clinical trial comparing dialectical behavior therapy and mentalization-based treatment in patients with borderline personality disorder? Psychol Med. 2019 Dec;49(16):2810-2811. doi: 10.1017/S0033291719001922. Epub 2019 Sep 19. No abstract available. PMID 31535604
- [Background] McGlashan TH, Grilo CM, Skodol AE, Gunderson JG, Shea MT, Morey LC, Zanarini MC, Stout RL. The Collaborative Longitudinal Personality Disorders Study: baseline Axis I/II and II/II diagnostic co-occurrence. Acta Psychiatr Scand. 2000 Oct;102(4):256-64. doi: 10.1034/j.1600-0447.2000.102004256.x. PMID 11089725
- [Background] McMurran M, Huband N, Overton E. Non-completion of personality disorder treatments: a systematic review of correlates, consequences, and interventions. Clin Psychol Rev. 2010 Apr;30(3):277-87. doi: 10.1016/j.cpr.2009.12.002. Epub 2009 Dec 13. PMID 20047783
- [Background] Meuldijk D, McCarthy A, Bourke ME, Grenyer BF. The value of psychological treatment for borderline personality disorder: Systematic review and cost offset analysis of economic evaluations. PLoS One. 2017 Mar 1;12(3):e0171592. doi: 10.1371/journal.pone.0171592. eCollection 2017. PMID 28249032
- [Background] Moran P, Rendu A, Jenkins R, Tylee A, Mann A. The impact of personality disorder in UK primary care: a 1-year follow-up of attenders. Psychol Med. 2001 Nov;31(8):1447-54. doi: 10.1017/s003329170105450z. PMID 11722159
- [Background] Karterud S, Pedersen G, Bjordal E, Brabrand J, Friis S, Haaseth O, Haavaldsen G, Irion T, Leirvag H, Torum E, Urnes O. Day treatment of patients with personality disorders: experiences from a Norwegian treatment research network. J Pers Disord. 2003 Jun;17(3):243-62. doi: 10.1521/pedi.17.3.243.22151. PMID 12839103
- [Background] Rohde C, Polcwiartek C, Correll CU, Nielsen J. Real-World Effectiveness of Clozapine for Borderline Personality Disorder: Results From a 2-Year Mirror-Image Study. J Pers Disord. 2018 Dec;32(6):823-837. doi: 10.1521/pedi_2017_31_328. Epub 2017 Nov 9. PMID 29120277
- [Background] Sansone RA, Farukhi S, Wiederman MW. Utilization of primary care physicians in borderline personality. Gen Hosp Psychiatry. 2011 Jul-Aug;33(4):343-6. doi: 10.1016/j.genhosppsych.2011.04.006. Epub 2011 May 20. PMID 21762830
- [Background] Soeteman DI, Hakkaart-van Roijen L, Verheul R, Busschbach JJ. The economic burden of personality disorders in mental health care. J Clin Psychiatry. 2008 Feb;69(2):259-65. doi: 10.4088/jcp.v69n0212. PMID 18363454
- [Background] Stoffers JM, Vollm BA, Rucker G, Timmer A, Huband N, Lieb K. Psychological therapies for people with borderline personality disorder. Cochrane Database Syst Rev. 2012 Aug 15;2012(8):CD005652. doi: 10.1002/14651858.CD005652.pub2. PMID 22895952
- [Background] Torgersen S, Kringlen E, Cramer V. The prevalence of personality disorders in a community sample. Arch Gen Psychiatry. 2001 Jun;58(6):590-6. doi: 10.1001/archpsyc.58.6.590. PMID 11386989
- [Background] Webb, D., & McMurran, M. (2009). A comparison of women who continue and discontinue treatment for borderline personality disorder. Personality and Mental Health, 3, 142-149.
- [Background] Zanarini MC, Frankenburg FR, Dubo ED, Sickel AE, Trikha A, Levin A, Reynolds V. Axis II comorbidity of borderline personality disorder. Compr Psychiatry. 1998 Sep-Oct;39(5):296-302. doi: 10.1016/s0010-440x(98)90038-4. PMID 9777282
- [Background] Zimmerman M, Chelminski I, Young D. The frequency of personality disorders in psychiatric patients. Psychiatr Clin North Am. 2008 Sep;31(3):405-20, vi. doi: 10.1016/j.psc.2008.03.015. PMID 18638643